CLINICAL TRIAL: NCT01607307
Title: Effect of Daikenchuto (TJ-100) on Intestinal Dysmotility and For the Prevention of Postoperative Paralytic Ileus in Patients Undergoing Pancreaticoduodenectomy: A Multicenter, Randomized, Placebo-Controlled Phase II Trial
Brief Title: Daikenchuto for Intestinal Dysmotility and Prevention of Postoperative Paralytic Ielus After Pancreaticoduodenectomy
Acronym: JAPAN-PD
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Wakayama Medical University (Other)
Collaborators: Epidemiological and Clinical Research Information Network (Other)
Responsible Party: Principal Investigator, Hiroki Yamaue, Professor, Wakayama Medical University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: JAPAN-PD; UMIN000007975 (Other: UMIN-CTR)
Record Dates: First submitted 2012-05-16; First posted 2012-05-30 (Estimated); Last update posted 2013-12-18 (Estimated); Status verified 2012-08

CONDITIONS: Paralytic Ileus
Keywords: daikenchuto; postoperative ileus; pancreaticoduodenectomy
MeSH Terms: conditions — Intestinal Pseudo-Obstruction

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Oral/enteral TJ-100 solution (Active Comparator): Oral/enteral TJ-100 solution
  Interventions: Drug: Oral/enteral TJ-100 solution
- Oral/enteral placebo solution (Placebo Comparator): Oral/enteral placebo solution
  Interventions: Drug: Oral/enteral placebo solution

INTERVENTIONS:
Drug: Oral/enteral TJ-100 solution — Oral TJ-100 solution (5 g tid, 15 g/day) given immediately before meals or every 8 h from preoperative day 3 to postoperative day 7 for 10 consecutive days. A diluent TJ-100 solution given immediately after surgery and on postoperative day 1 via Argyle enteral feeding tube (10 Fr), which terminates in the jejunum to prevent aspiration pneumonia.
  Other Names: A
  Arms: Oral/enteral TJ-100 solution
Drug: Oral/enteral placebo solution — Oral placebo solution (5 g tid, 15 g/day) given immediately before meals or every 8 h from preoperative day 3 to postoperative day 7 for 10 consecutive days. A diluent placebo solution given immediately after surgery and on postoperative day 1 via Argyle enteral feeding tube (10 Fr), which terminates in the jejunum to prevent aspiration pneumonia.
  Other Names: B
  Arms: Oral/enteral placebo solution

SUMMARY:
A multicenter randomized-controlled trial of daikenchuto (TJ-100), a traditional Japanese herbal medicine (Kampo), to investigate its effect on intestinal dysmotility and for the prevention of postoperative paralytic ileus.

DETAILED DESCRIPTION:
Daikenchuto (TJ-100), a traditional Japanese herbal medicine, is used for prevention and treatment of postoperative ileus. TJ-100 extract powder (Tsumura & Co., Tokyo, Japan) is manufactured as an aqueous extract containing 2.2 % Japanese pepper, 5.6 % processed ginger, 3.3 % ginseng, and 88.9 % maltose syrup powder. A recent randomized, parallel-group, double-blind, placebo-controlled, dose-response trial demonstrated that TJ-100 accelerates colonic transit time, particularly in the ascending colon. Given its potential actions in the intestinal tract, it seems reasonable to postulate that TJ-100 may play a role in improving and preventing bowel dysmotility. This study was designed to investigate the effect of TJ-100 on intestinal dysmotility and for the prevention of postoperative paralytic ileus in patients undergoing pancreaticoduodenectomy.

The primary endpoint is the incidence of postoperative paralytic ileus. Secondary endpoints are QOL assessment by the Gastrointestinal Symptom Rating Scale (GSRS) Score (Japanese Version) and visual analogue scale, the change in ratio of abdominal circumference, the incidence of postoperative complications, the length of hospital day, and the incidence of surgical site infection. Two hundred patients are required for the study (100 patients per group).

ELIGIBILITY:
Inclusion Criteria:

* Patients with periampullary tumors (extrahepatic bile duct tumor, tumors of ampulla of Vater and duodenal tumor) and pancreatic tumors (pancreatic cancer, intraductal papillary mucinous neoplasm of the pancreas, pancreatic endocrine tumor and pancreatic neuroendocrine tumor) of the head of the pancreas who are scheduled to undergo PD.
* Age of at least 20 years old at the time of registration.
* All patients provided written informed consent before initiation of study-related procedures.

Exclusion Criteria:

* Clinically problematic cardiac disease.
* Liver cirrhosis or active hepatitis.
* Severe pulmonary disease (interstitial pneumonia, pulmonary fibrosis, pulmonary emphysema etc.).
* Chronic renal failure requiring hemodialysis.
* Other malignant disease that can influence the adverse effect.
* Patients with tumors requiring resection of colon.
* Patients who are expected to have severe intra-abdominal adhesion due to past surgical history or past peritonitis history.
* Patients who had used gastrointestinal prokinetic medication, antipsychotic medication or antidepressants.
* Patients who had used Japanese herbal (Kampo) medicines within 4 weeks before registration.
* Pregnant or lactating women.
* Any other medical condition that makes the patient unsuitable for inclusion in the study according to the opinion of the investigator.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 220 (Estimated)
Dates: Start 2012-08; Primary Completion 2013-12 (Actual); Study Completion 2016-08 (Estimated)

PRIMARY OUTCOMES:
Incidence of postoperative paralytic ileus (including the duration of paralysis) | 72 hours
  Delayed passage of first flatus for 72 hours (3.0 days) after surgery, or a postoperative condition that requires an intervention for the ileus. Every 12 hours is counted as 0.5 postoperative day and every 24 hours as 1.0 postoperative day.
The duration until the first flatus after surgery. | 14 days
  The first passages of flatus will be confirmed by patients themselves and they will inform it to the medical staffs.

SECONDARY OUTCOMES:
QOL assessment by the Gastrointestinal Symptom Rating Scale (GSRS) Score (Japanese Version) | 7 days
  QOL assessment by the Gastrointestinal Symptom Rating Scale (GSRS) Score (Japanese Version) on postoperative day 7.
Abdominal pain and abdominal distention scores on the Visual Analogue Scale. | 3 days
  Abdominal pain and abdominal distention scores on the Visual Analogue Scale on postoperative day 3.
The change ratio of abdominal circumference. | 3 days
  The change ratio of abdominal circumference on postoperative day 3 and operative day just after surgery
The incidence of postoperative complication. | 14 days
  The incidence of postoperative complication based on Dindo's classification.
The length of postoperative hospital day. | 30 days
  Patients were discharged only when they fulfilled the criteria as follows: a return to preoperative activities of daily living, no deep-site infections, normal laboratory data, no drains, and the possibility for oral nutrition above the basal metabolism.
The incidence of surgical site infection. | 30 days
  Intra-abdominal abscess was defined as intra-abdominal fluid collection with positive cultures identified by ultrasonography or computed tomography associated with persistent fever and elevations of white blood cell counts.
The long term incidence of postoperative ileus after surgery. | 2 years
  The follow-up investigation of the long term incidence of postoperative ileus is scheduled in two years after surgery.

CONTACTS AND LOCATIONS:
Overall Officials: Hiroki Yamaue, M.D., Ph.D., Principal Investigator — Second Department of Surgery, Wakayama Medical University
Locations (5):
- Japan (5):
  - Nagoya University, Nagoya, Aichi-ken
  - Hiroshima University, Hiroshima, Hiroshima
  - Osaka University, Suita, Osaka
  - Shizuoka Cancer Center Hospital, Shizuoka, Shizuoka
  - Wakayama Medical University, Wakayama, Wakayama

REFERENCES:
- [Derived] Maeda H, Okada KI, Fujii T, Oba MS, Kawai M, Hirono S, Kodera Y, Sho M, Akahori T, Shimizu Y, Ambo Y, Kondo N, Murakami Y, Ohuchida J, Eguchi H, Nagano H, Sakamoto J, Yamaue H. Transition of serum cytokines following pancreaticoduodenectomy: A subsidiary study of JAPAN-PD. Oncol Lett. 2018 Nov;16(5):6847-6853. doi: 10.3892/ol.2018.9422. Epub 2018 Sep 7. PMID 30333892
- [Derived] Okada K, Kawai M, Hirono S, Fujii T, Kodera Y, Sho M, Nakajima Y, Satoi S, Kwon AH, Shimizu Y, Ambo Y, Kondo N, Murakami Y, Ohuchida J, Eguchi H, Nagano H, Oba MS, Morita S, Sakamoto J, Yamaue H; JAPAN-PD Investigators. Evaluation of the efficacy of daikenchuto (TJ -100) for the prevention of paralytic ileus after pancreaticoduodenectomy: A multicenter, double-blind, randomized, placebo-controlled trial. Surgery. 2016 May;159(5):1333-41. doi: 10.1016/j.surg.2015.11.019. Epub 2015 Dec 31. PMID 26747224